CLINICAL TRIAL: NCT06153225
Title: Amino Acid Concentrations in Serum After Intake of Plant Based Protein Sources
Brief Title: Amino Acid Concentrations in Serum After Intake of Different Protein Sources
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nutricia Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SBB22R&40716
Record Dates: First submitted 2023-04-07; First posted 2023-12-01 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-11

CONDITIONS: Postprandial Amino Acid Concentrations in Healthy Adults
Keywords: Postprandial; Healthy individuals; Amino acid; Bioavailability; Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub study 1 (Experimental): All subjects will receive 4 study products (300ml each) on 4 different visits in a randomized order. In total in both arms combined, 7 products will be tested.
  Interventions: Dietary Supplement: Protein products
- Sub study 2 (Experimental): All subjects will receive 4 study products (300ml each) on 4 different visits a randomized order. In total in both arms combined, 7 products will be tested.
  Interventions: Dietary Supplement: Protein products

INTERVENTIONS:
Dietary Supplement: Protein products — In total 4 protein products will be tested containing a single or mixture of plant and dairy protein sources in a randomized order

SUMMARY:
This study assesses the amino acid concentrations in subject serum after intake of different types of proteins. The study is divided in two consecutive sub-studies. Subjects will be asked to ingest a specific protein blend each visit in a randomized order, after which blood will be drawn on 14 different time points. At least 48 hours will be kept between each visit, and the subjects receive a follow up call within 4-14 days after visit 4.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 70 years
2. Body Mass Index (BMI) ≥ 18.5 and ≤ 27.0 kg/m2
3. Written informed consent
4. Willingness and ability to comply with the protocol
5. Judged by the Investigator to be in good health

Exclusion Criteria:

1. Any gastrointestinal (GI) disease or surgery that may interfere with GI function and/or protein metabolism, including but not limited to phenylketonuria, pancreatitis, short bowel syndrome, celiac disease, Crohn's disease, in the opinion of the Investigator
2. Known renal or hepatic diseases that may interfere with protein metabolism, including but not limited to acute hepatitis, chronic liver disease, nephritis, cystinuria, chronic kidney disease, in the opinion of the Investigator
3. Use of systemic antibiotics, anticonvulsants, prokinetics, antacids, medication influencing gastric acid production, systemic anticoagulants, systemic corticosteroids, laxatives, growth hormone, testosterone, immunosuppressants or insulin within the past 3 weeks prior to screening
4. Allergy to soy, pea and/or cow's milk protein
5. Adherence to a weight loss program
6. Current eating disorder, e.g. anorexia nervosa or bulimia
7. Known pregnancy and/or lactation
8. Current smoking or stopped smoking for < 1 month prior to screening (except for incidental smoking of ≤ 3 cigarettes/cigars/pipes per week on average in the last month prior to screening)
9. Average alcohol use of > 21 glasses per week for men or > 14 glasses per week for women (on average during the last 6 months prior to screening)
10. Drug or medicine abuse in opinion of the investigator
11. Any known bleeding disorder
12. Known difficulties with placement of and/or blood drawings from a cannula
13. Active participation in any other study with investigational or marketed products concomitantly or within 4 weeks prior to screening
14. Major medical or major surgical event requiring hospitalization within the preceding 3 months and/or scheduled in the period of study participation
15. Investigator's uncertainty about the willingness or ability of the subject to comply with the protocol requirements
16. Employees of Nutricia Research and/or their family members or relatives

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-04-15 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Amino Acid concentration in blood | 240 minutes after dietary protein ingestion
  Relative content of amino acids in dietary protein and relative amount of amino acids appearing in the blood for the 4 hour period after the ingestion of different products [μmol]

SECONDARY OUTCOMES:
Individual Amino Acid concentration in blood | 240 minutes after dietary protein ingestion
  Postprandial serum concentrations of individual amino acids [μmol/L]

CONTACTS AND LOCATIONS:
Locations (1):
- NCRU, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No